CLINICAL TRIAL: NCT06359938
Title: Respiratory Sinus Arrhythmia Pacing Post-CABG Surgery in Patients With HFrEF
Brief Title: Respiratory Sinus Arrhythmia (RSA) Pacing Post-CABG Surgery in Patients With HFrEF
Acronym: RSA-PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceryx Medical Ltd (Industry)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cer22/01
Record Dates: First submitted 2023-03-14; First posted 2024-04-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; respiratory sinus arrhythmia; pacemaker
MeSH Terms: conditions — Heart Failure; Arrhythmia, Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial pacing with respiratory sinus arrhythmia (RSA) variability (Experimental): The experimental arm is atrial pacing with additional respiratory sinus arrhythmia (RSA) modulation following coronary artery bypass graft (CABG) surgery. Pacing impulses will be grouped together during inspiration, such that heart rate (HR) will increase by approximately 6 bpm above median during inspiration, and decrease by around 6 bpm below median during expiration. Five pacing rates will be used to accommodate a range of patients' intrinsic HR.
  Pacing will be initiated after randomisation, after the patient is removed from ventilator support (Pacing Day 1, PD1). This is usually the day after surgery. Pacing will continue until the patient is ready for discharge or there is a clinical decision to stop pacing and remove the leads (whichever is soonest).
  Pacing is delivered by a PACE204 pacemaker (Osypka Medical AG) modulated to respiratory phase by a Ceryx device (intervention)
  Interventions: Device: Atrial pacing with respiratory sinus arrhythmia (RSA) variability
- Monotonic atrial pacing (Active Comparator): The control arm is standard monotonic right atrial pacing at the relevant median rate following coronary artery bypass graft (CABG) surgery. Pacing will be initiated after randomisation, after the patient is removed from ventilator support (Pacing Day 1, PD1). This is usually the day after surgery. Pacing will continue until the patient is ready for discharge or there is a clinical decision to stop pacing and remove the leads (whichever is soonest).
  Pacing is delivered by a PACE204 pacemaker (Osypka Medical AG) delivering standard monotonic right atrial pacing.
  Interventions: Device: Monotonic right atrial overdrive pacing

INTERVENTIONS:
Device: Atrial pacing with respiratory sinus arrhythmia (RSA) variability — The intervention in this study is a modification of the pacing output from a standard external pacemaker such that it will approximate the RSA variation found in healthy subjects. A pacemaker (PACE204, Osypka Medical AG), similar to those currently in common use in post-CABG patients, will be adapted to receive an additional input signal based on the respiratory signal (Ceryx device). The respiration signal will be combined with the ECG signal to determine the appropriate pacing interval. The pacing impulse will be delivered by the pacemaker unit.
  Other Names: Modified temporary external pacemaker (Osypka) with additional pacing RSA module (Ceryx box)
  Arms: Atrial pacing with respiratory sinus arrhythmia (RSA) variability
Device: Monotonic right atrial overdrive pacing — Pacing is delivered by a PACE204 pacemaker (Osypka Medical AG) delivering standard monotonic right atrial pacing
  Other Names: PACE204 pacemaker (Osypka Medical AG) delivering standard monotonic right atrial pacing
  Arms: Monotonic atrial pacing

SUMMARY:
The goal of this clinical trial is to test a new type of pacemaker in heart failure patients following a heart bypass operation. The new pacemaker restores respiratory sinus arrhythmia which is a natural pattern where the heart rate increases when the participants breathe in and slows down when participants breathe out.

The main questions the trial aims to answer are:

* Is the new type of pacemaker safe?
* Does the new type of pacemaker improve how patients' hearts work (also known as cardiac output)?

Participants will have a range of tests before their operation and during their recovery in hospital while participants have the new type of pacemaker in place, and will be monitored very closely. Participants will also receive a phone call 1 month after their surgery. Researchers will compare the new type of heart pacing against standard treatment to see if it is as safe, and if it is any better for patients.

DETAILED DESCRIPTION:
This is a first-in-human (FIH) clinical investigation of a modification of an existing medical device. It will be a comparative, multicentre, randomised controlled trial (RCT) design. RSA modulated atrial pacing will be compared against monotonic atrial pacing in patients with HFrEF who have had CABG surgery.

The purpose of this clinical investigation is to explore the risk/benefit profile of the use of RSA pacing in patients with HFrEF following CABG. Based on the prior animal models the investigators hypothesise an improvement in cardiac function over several days of RSA pacing, with no increase in risk compared to typical pacemaker use.

Primary hypothesis - Atrial pacing with additional RSA variability (for up to 10 days) is feasible and safe in patients with heart failure and reduced ejection fraction. The primary outcome is measuring arrhythmia episodes.

Secondary hypothesis - Atrial pacing with additional RSA variability improves cardiac function in patients with heart failure and reduced ejection fraction following CABG surgery. The secondary outcomes is measuring cardiac function, cardiac output, apnoea episodes.

Respiratory sinus arrhythmia is part of normal physiology and RSA pacing is looking to restore this. In heart failure, RSA is severely reduced. Therefore the investigators have identified that, post-CABG surgery patients with heart failure and reduced ejection fraction are the ideal candidates for this study. Following surgery it is standard of care for a surgeon to leave temporary pacing wires attached to the heart as a precaution and it is not uncommon to leave them in for 10 days or longer. Hence, these temporary wires can be used to deliver RSA pacing. Adjusting pacing rates is common in both implanted or temporary pacemakers.

Potential patients awaiting CABG surgery with heart failure with reduced ejection fraction will be identified using two routes - inpatients and outpatients.

The investigators would randomly allocate patients to either the RSA external pacemaker box or the normal external pacemaker for a maximum of 10 days. Patients will be connected to nasal prongs to monitor their respiration and in the RSA group, this signal will be fed to the external pacemaker to deliver RSA pacing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 22 years) selected for isolated, on-pump coronary artery bypass graft (CABG)
* Established diagnosis of heart failure with reduced ejection fraction (HFrEF).
* Elective or urgent admission routes
* Echocardiography assessment of left ventricular ejection fraction (EF) of 20%-40% (within 1 month of planned surgery)
* Sinus rhythm
* Any number of coronary vessels replaced. Must include left anterior descending artery.
* Able to provide written informed consent

Exclusion Criteria:

* Requirement for concurrent valve replacement surgery.
* Off-pump CABG.
* Emergency CABG
* History of paroxysmal or permanent atrial fibrillation or flutter
* History of atrioventricular-node dependent tachycardia
* Patients lacking capacity to consent
* Patient testing positive for Covid-19 within 14 days of intended CABG (PCR or lateral flow test)
* Intrinsic resting heart rate > 100bpm
* Pregnancy
* Implanted pacemaker or defibrillator
* Failure to obtain Uscom signals

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of arrhythmia episodes per patient during pacing | From start of pacing to end of pacing
  Any episode of arrhythmia, captured on an ECG between the initiation of pacing (Pacing Day 1) and the post-pacing visit (Day 7 - Post-discharge form hospital ), and lasting 30 seconds or longer, will be recorded. Anonymised ECG extracts will be reviewed by two cardiologists to identify the type of arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Yousef, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Cardiff & Vale University Health Board, Cardiff, United Kingdom